CLINICAL TRIAL: NCT06353750
Title: Exploring Intramyocellular Magnesium Augmentation: Implications for Myocardial and Skeletal Muscle Metabolism in Individuals With Heart Failure With Preserved Ejection Fraction
Brief Title: Intracellular Magnesium and Heart Failure
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: British Heart Foundation (Other); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 331039
Record Dates: First submitted 2024-04-02; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Hypomagnesemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals with heart failure with preserved ejection fraction (HFpEF): * Clinical diagnosis of HFpEF
  * HFA-PEFF score ≥ 5
  Interventions: Other: Magnesium supplement
- Healthy controls: * HFA-PEFF < 3
  * No known diagnosis of heart failure
  Interventions: Other: Magnesium supplement
- Matched controls: * HFA-PEFF < 3
  * No known diagnosis of heart failure
  * Age and sex-matched individuals to the HFpEF cohort
  Interventions: Other: Magnesium supplement

INTERVENTIONS:
Other: Magnesium supplement — Intravenous magnesium supplement (10mmol).

SUMMARY:
Low magnesium levels are surprisingly common in those with a heart condition known as HFpEF, where the heart pumps well but is too rigid to fill properly with blood. While routine blood tests can check magnesium levels, they don't tell us how much magnesium is actually inside the heart and muscle cells, where it's vital for energy and overall function. Our research aims to get a clearer picture by looking directly at the magnesium inside these cells and understanding its role in the body's energy production and usage. We're also interested in how magnesium levels affect symptoms and the body's handling of sugar. We're using advanced medical imaging techniques, like heart magnetic resonance imaging (MRI) and other heart and muscle function tests, at rest and when the heart is working hard to help answer these questions. We'll compare the magnesium levels inside the cells before and after giving a supplement of magnesium to see if this can make a difference in how the heart and muscles work.

DETAILED DESCRIPTION:
Hypomagnesaemia is prevalent among patients suffering from heart failure with preserved ejection fraction (HFpEF), and in those with predisposing risk factors such as obesity and diabetes. The intricate link between hypomagnesaemia and the pathophysiological processes of HFpEF remains to be fully elucidated. However, its notable prevalence suggests a significant role in the onset and advancement of the disease. Serum magnesium (S-Mg) is commonly used to evaluate Mg status, however, it does not accurately reflect true intracellular Mg concentrations ([Mg2+]i), where this essential ion exerts its beneficial effects. Thus, previous literature lacks a thorough evaluation of [Mg2+]i in HFpEF, and specifically the potential impact of Mg replete physiology.

The research hypothesis is that [Mg2+]i is related to myocardial and skeletal muscle (SM) energetics and performance in patients with HFpEF. The study aims to explore the role of [Mg2+]i at a functional and cellular level in cardiac and SM, symptomatology, and insulin sensitivity; comparing a HFpEF population with healthy and matched controls.

Using the chemical shift difference in the resonance frequencies of the α- and β- phosphate resonances in magnetic resonance spectroscopy (MRS), [Mg2+]i will be measured, comparing it to S-Mg. Blood samples for cardiac biomarkers, electrolytes, and markers of HFpEF risk factors (such as lipid profile, HbA1C and TSH) will be taken and a calf leg raise performed. Advanced imaging techniques at rest and stress including cardiac magnetic resonance imaging (CMR), MRS and echocardiography will be performed. MRS measurements include cellular energetics (Phosphocreatine [PCr]/ATP), rate of myocardial ATP delivery (CK flux and KfCK) and skeletal muscle energetics (PCr recovery Tau). At two time points post-Mg augmentation (immediate and delayed [7-15 days]), investigations will be repeated.

This study aspires to quantify [Mg2+]i in the HFpEF population compared with healthy and matched controls, juxtapose its levels with S-Mg, and examine its significance in the pathophysiology, functional and cellular performance, and symptom presentation of HFpEF. The study aims to recruit 45 individuals with HFpEF, 20 healthy controls and 20 age-and sex-matched individuals over a 2-year period.

ELIGIBILITY:
General Inclusion Criteria

* Participant is willing and able to give informed consent for participation in the study.
* Participant aged at least 18 years old.

6.2.2 Additional inclusion criteria for participants in the HFpEF arm

* Clinical diagnosis of HFpEF
* HFA-PEFF score ≥ 5

6.2.3 Additional inclusion criteria for participants in the healthy and matched control arm

* HFA-PEFF < 3
* No known diagnosis of heart failure

6.3 Exclusion criteria

* Participant is unwilling or unable to give informed consent
* Any impediment to communication which, in the opinion of the investigator, might prevent the investigator communicating effectively with the patient during the study which could cause a safety or reliability concern.
* Any other condition which, in the opinion of the investigator, might affect the safety of the participant or reduce the reliability of the study results
* Involvement in any other research project where the procedures would affect the outcomes of this study.
* Individuals with NYHA class IV symptoms
* Known ischaemic heart disease, ICD, or CRT in situ.
* Individuals on oral magnesium supplementation
* Insulin dependent diabetes
* Standard contraindications to magnetic resonance imaging (MRI), (Metal clips or metallic foreign body, prior injury to the eye involving fragments of metal, prior shrapnel injuries, any other metallic or electronic implants affected by the magnetic field, history of severe claustrophobia, history of chronic kidneys disease, egg, or soya allergy)
* Heart transplant recipient
* Cardiomyopathy from infiltrative or storage diseases, muscular dystrophies, or with reversible causes, hypertrophic cardiomyopathy
* Moderate or greater valvular heart disease
* Acute HF requiring iv diuretics, inotropes, vasodilators, or hospitalisation within 6 weeks of screening
* BMI>40kg/m2 (due to MRS sensitivity).
* Pregnancy (due to magnesium infusion).
* Chronic kidney disease stage 4/5 (due to contrast injection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study investigators will contact those people who have participated in other ethically approved studies conducted at the research centre and have consented for their contact details to be retained in order to be contacted to take part in other research.
  Patients attending outpatient heart failure clinics will be identified by their routine clinical care team. Patients attending for clinical cardiac imaging as part of their routine care who indicate on their consent form that they are happy to take part in research will be identified by their routine clinical team.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
Myocardial/ skeletal muscle metabolism and energetics at rest and stress. | 7-15 days
  Measuring myocardial metabolism (PCr/ATP, CK flux and KfCK, PDH flux), and skeletal muscle metabolism (PCr recovery Tau) at rest and stress. Measurements at three time points (pre-Mg infusion, immediately post and delayed (7-15 days) after Mg infusion, comparing HFpEF population with healthy and matched controls.

SECONDARY OUTCOMES:
Serum versus intracellular magnesium concentration | 7-15 days
  Comparing serum magnesium with intracellular magnesium concentrations using MRS, at all time points (pre-Mg infusion, and post (immediately and 7-15 days after) Mg infusion).
Cardiac function | 7-15 days
  Comparing systolic and diastolic function (echocardiography) at rest and exercise at the three time points (pre-Mg infusion, immediately post and delayed (7-15 days) after Mg infusion), and assessing if [Mg2+] has a stronger correlation with cardiac function than serum Mg2+.
Skeletal muscle performance | 7-15 days
  Comparing Calf raise test at the three time points (pre-Mg infusion, immediately post and delayed (7-15 days) after Mg infusion), and assessing if [Mg2+] has a stronger correlation with test performance than serum Mg2+.
Symptoms | 7-15 days
  To assess if Mg2+ infusion affects perceived exercise tolerance (NYHA class and symptom questionnaire) at 2 time points (pre-Mg infusion, and 7-15 days post-Mg infusion).
Insulin sensitivity | 7-15 days
  To assess if Mg2+ infusion affects a HOMA-IR score (based on fasted serum glucose and insulin levels).
  To assess if Mg2+ infusion affects a HOMA-IR score (based on fasted serum glucose and insulin levels).
  To assess if Mg2+ infusion affects a HOMA-IR score (based on fasted serum glucose and insulin levels).
  To assess if Mg2+ infusion affects a HOMA-IR score (based on fasted serum glucose and insulin levels), comparing 2 time points (pre-Mg infusion, and 7-15 days post-Mg infusion).

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford Centre for Magnetic Resonance (OCMR), Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No